CLINICAL TRIAL: NCT06763003
Title: Feasibility Randomised Controlled Trial of Intensive Music Therapy on Cognitive Function in Subacute Stroke Rehabilitation in Malaysia
Brief Title: Intensive Music Therapy on Cognitive Function in Subacute Stroke Rehabilitation in Malaysia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr. Beh Wen Fen, Dr, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Intensive MT
Record Dates: First submitted 2024-12-22; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Rehabilitation; Cognition; Stroke; Attention
Keywords: Music therapy; randomised controlled trial; rehabilitation; stroke; cognition; attention
MeSH Terms: conditions — Stroke | interventions — Music Therapy; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant, care provider, investigator and outcome assessor will be evaluated by different disciplines.
  1. Participant - ramdomised by principal investigator
  2. care provider - music therapist
  3. Investigator - rehabilitation specialist
  4. outcome assessor - neuropsychologist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care group (Active Comparator): In the control group, participants will receive the standard neurorehabilitation program prescribed by the rehabilitation team, without the addition of music therapy. This will provide a baseline to compare outcomes with the intervention group and evaluate the feasibility and preliminary effects of the music therapy intervention. The usual cognitive rehabilitation program during the subacute stroke period focuses on restoring cognitive abilities such as attention, memory, executive functions, and communication. The control group's daily rehabilitation sessions will last for 45 minutes, mirroring the music therapy group's session duration, ensuring a fair comparison of outcomes across both groups. This comparison will help assess the unique contributions of music therapy on cognitive functions like attention, memory, and executive functions in stroke patients.
  Interventions: Other: Standard Care (in control arm)
- Music Therapy Group (Experimental): The music therapy session described follows a structured and engaging approach, aimed at enhancing the patient's cognitive skills during neurorehabilitation. Here's a summary of the session components: Relaxation Phase, Song Selection, Instrument Selection and Familiarization, Rhythmic Training, Progression and Adjustment, Session Frequency and Customization. This individualized approach aims to enhance patient engagement and recovery by integrating music, rhythm, and therapeutic interaction into the neurorehabilitation process.
  Interventions: Other: Music Therapy

INTERVENTIONS:
Other: Music Therapy — The music therapy session described follows a structured and engaging approach, aimed at enhancing the patient's cognitive skills during neurorehabilitation. Here's a summary of the session components: Relaxation Phase, Song Selection, Instrument Selection and Familiarization, Rhythmic Training, Progression and Adjustment, Session Frequency and Customization. This individualized approach aims to enhance patient engagement and recovery by integrating music, rhythm, and therapeutic interaction into the neurorehabilitation process.
  Arms: Music Therapy Group
Other: Standard Care (in control arm) — In the control group, participants will receive the standard neurorehabilitation program prescribed by the rehabilitation team, without the addition of music therapy. This will provide a baseline to compare outcomes with the intervention group and evaluate the feasibility and preliminary effects of the music therapy intervention. The usual cognitive rehabilitation program during the subacute stroke period focuses on restoring cognitive abilities such as attention, memory, executive functions, and communication. The control group's daily rehabilitation sessions will last for 45 minutes, mirroring the music therapy group's session duration, ensuring a fair comparison of outcomes across both groups. This comparison will help assess the unique contributions of music therapy on cognitive functions like attention, memory, and executive functions in stroke patients.
  Arms: Standard Care group

SUMMARY:
The purpose of this study is to explore whether intensive music therapy can help improve cognitive functions like memory, attention, and decision-making skills in stroke patients who are undergoing rehabilitation.

This is a feasibility study, meaning it's also designed to see how practical it is to include music therapy as part of stroke rehabilitation. The investigators want to learn how well patients can participate in and stick with this type of therapy, and whether it fits well with other treatments that stroke patients usually receive. By understanding this, the investigators can assess the resources, staff training, and planning needed for music therapy to be part of stroke recovery in the future.

The study will also help the investigators estimate the effects of music therapy, which will be used to design a larger, more detailed study in the future.

DETAILED DESCRIPTION:
This study will be a feasibility randomised controlled trial (RCT) in one centre, with two parallel groups: an intervention group receiving intensive music therapy in addition to standard neurorehabilitation, and a control group receiving only standard neurorehabilitation. A certified music therapist will conduct the intervention and a trained assessor will evaluate the outcome. The assessor is blinded to the patients' allocation group and will evaluate the cognitive outcomes at baseline, at two weeks (after 8 sessions) and at 1 month post intervention. All patients whoare admitted to the rehabilitation ward for stroke rehabilitation will be screened and approached. Informed consent will be obtained from eligible patients before randomisation. To ensure that there are exactly 15 patients in both the control and intervention groups, block randomization will be used using a random number generator. After randomization, the group assignments will be kept in a password-protected file that only the study coordinator can access. The assessor will not have access to this information because the patients will be labelled with anonymous codes that do not reveal whether they are in the control or intervention group. The assessor will only know the code, not the group assignment, ensuring unbiased evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ischemic or haemorrhagic stroke confirmed by CT scan
* Duration of stroke within the first 3 months
* Aged 18 - 75 years old
* Ability to provide informed consent
* Understands Bahasa Melayu or English with basic communication abilities to follow instructions during therapy sessions
* Mild to moderate cognitive impairments with MoCA score of 10-25.

Exclusion Criteria:

* Severe aphasia
* Significant uncorrected hearing or visual impairments preventing engagement in music therapy.
* Severe or unstable medical conditions (e.g., uncontrolled hypertension or diabetes).
* Medications that significantly impair cognition or motor function (e.g., high dose sedatives).
* History of neurological diseases other than stroke (eg, Parkinson's disease).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | This will be assessed at baseline, after completion of 8 sessions, an average of 2 weeks and also at 1 month after completion.
  is noteworthy for being greater sensitivity than the other test and can detect more mild deficits
Trail Making Test (TMT) | This will be assessed at baseline, after completion of 8 sessions, an average of 2 weeks and also at 1 month after completion.
  is easy to understand, and has a short administration which assesses visuoperceptual tracking, processing speed, divided attention, and cognitive flexibility.
Digit Span (Forward and Backward) | This will be assessed at baseline, after completion of 8 sessions, an average of 2 weeks and also at 1 month after completion.
  is easy to implement, requires minimal training needs, and measures selective attention and cognitive interference
Clock Drawing Test (CDT) | This will be assessed at baseline, after completion of 8 sessions, an average of 2 weeks and also at 1 month after completion.
  is a screening test for cognitive dysfunction secondary to dementia, delirium, or a range of neurological and psychiatric illnesses

IPD SHARING:
Plan to Share IPD: Undecided
For confidentiality purposes.

REFERENCES:
- [Result] Fang R, Ye S, Huangfu J, Calimag DP. Music therapy is a potential intervention for cognition of Alzheimer's Disease: a mini-review. Transl Neurodegener. 2017 Jan 25;6:2. doi: 10.1186/s40035-017-0073-9. eCollection 2017. PMID 28149509
- [Result] Koo SC, Moon BC, Kim JK, Kim CY, Sung SJ, Kim MC, Cho MJ, Cheong YH. OsBWMK1 mediates SA-dependent defense responses by activating the transcription factor OsWRKY33. Biochem Biophys Res Commun. 2009 Sep 18;387(2):365-70. doi: 10.1016/j.bbrc.2009.07.026. Epub 2009 Jul 14. PMID 19607808
- [Result] Alluri V, Toiviainen P, Jaaskelainen IP, Glerean E, Sams M, Brattico E. Large-scale brain networks emerge from dynamic processing of musical timbre, key and rhythm. Neuroimage. 2012 Feb 15;59(4):3677-89. doi: 10.1016/j.neuroimage.2011.11.019. Epub 2011 Nov 12. PMID 22116038
- [Result] Thaut, M. H. (2010). Neurologic Music Therapy in cognitive rehabilitation. Music Perception, 27(4), 281-285.
- [Result] Thaut MH, Gardiner JC, Holmberg D, Horwitz J, Kent L, Andrews G, Donelan B, McIntosh GR. Neurologic music therapy improves executive function and emotional adjustment in traumatic brain injury rehabilitation. Ann N Y Acad Sci. 2009 Jul;1169:406-16. doi: 10.1111/j.1749-6632.2009.04585.x. PMID 19673815

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/03/NCT06763003/Prot_ICF_000.pdf